CLINICAL TRIAL: NCT05679011
Title: Analysis of Optimal Acceleration/Deceleration Distance in Gait Speed Tests With Motion Capture System in Chronic Post-stroke. Cross-sectional Study
Brief Title: Analysis Acceleration/Deceleration Distance Gait Speed Tests in Stroke Survivors
Acronym: Walk-test
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, Senior lecturer, Universitat Internacional de Catalunya
Other Study IDs: Gait speed optimal distance
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Chronic Stroke
Keywords: gait speed; comfortable gait speed; acceleration distance; walking test; 10mWT; 6mWT; fast speed; 6 meters walk test; 4 meters walk test; deceleration distance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 4 and 6 meters walking test — A 10-meter and other 6-meter flats pathways were identified. Two-meter are provided for the acceleration zone and two-meter for deceleration for 6-meter walk test. One meter to acceleration and another to deceleration for 4-meter walk test. The participants are randomly to perform 3-time to comfortable speed and 3-time faster speed for 4-meter and 6-meter.

SUMMARY:
Introduction: Gait speed is currently used to predict the future functional status of the patient or to evaluate the improvements produced by different neurorehabilitation treatments. There is no common agreement among researchers and clinicians as to the optimal distance required to accelerate and decelerate in walking tests (4-meter and 6-meter timed) in people in the chronic phase of stroke.

Objectives: The main objective is to analyze what is the optimal distance to accelerate and decelerate in the 4-meter walk test (4mWT) and 6-meter walk test (6mWT) at comfortable and fast speed with optical motion capture for chronic stroke survivors (> 6 months).

The secondary objective is to evaluate whether the mean gait speed taken by stopwatch is comparable to optical motion capture system Optitrack for the 4mWT and the 6mWT for a correct measurement of gait at comfortable and fast speed in in chronic stroke survivors.

Methods: A cross-sectional observational study is performed. The walking speed is measured using the OptiTrack optical motion capture system consisting of 8 PrimeX 13 cameras and Motive 2.0 capture and analysis software (Natural Point Inc. Corvallis OR USA).The patient ware 8 markers sensors applied to different parts of the body. The two tests are performed first at a comfortable gait and second at the fastest gait that the patient can safely perform. There were 3 repetitions for each of the tests. The individuals are randomized to start with either the 6mWT or the 4mWT test. All tests are performed on the same day.

Discussion: This study will shed light on what is the optimal distance required for acceleration and deceleration phases on the 6mWT and 4mWT walking tests at comfortable and fast speed.

DETAILED DESCRIPTION:
Gait disorder is a common clinical problem after stroke and is among the prevalent physical limitations contributing to stroke-related disability that impacts performance of activities of daily(1). Gait disturbances in patients with stroke are caused by weakness (paresis or paralysis), abnormal tone in the limbs or trunk, or by disturbances in the sensory-motor system or central control mechanisms.(2) Therefore, gait recovery is a major objective in the rehabilitation program in stroke survivors.(3) Walking speed is considered to be the sixth vital sign (4). Clinical practice guidelines worldwide recommend using reliable and valid tools to assess walking in stroke rehabilitation.(5,6) The 10 meter walk test at comfortable speed is widely recommended to reflect a walking speed. (7) However, there are many different distances to accelerate and decelerate.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors in chronic phase > 6 months
* Have preserved cognitive ability: Achieve a score equal to or greater than 25 points on the Montreal Cognitive Assessment test.
* Have the ability to walk on a flat surface of at least 10 meters, with or without aid.

Exclusion Criteria:

A history of lower extremities injury or surgery

* A history of botulinum injection within 3 months
* A history of inflammatory arthritis
* A history of inflammatory myopathy or peripheral nervous disease
* A history of other neurological disease as a Parkinson, spinal cord etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors in chronic phase > 6 months
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Acceleration/deceleration distance for 6mWT at comfortable speed | 15 minutes
  Distance time that an individual needs to reach their average gait speed. Examinees are timed once the first foot passes the acceleration path; the time is stopped once the first foot enters the deceleration path.
Acceleration/deceleration distance for 4mWT at comfortable speed | 15 minutes
  Distance time that an individual needs to reach their average gait speed. Examinees are timed once the first foot passes the acceleration path; the time is stopped once the first foot enters the deceleration path.
Acceleration/deceleration distance for 6mWT at fast speed | 15 minutes
  Distance time that an individual needs to reach their average gait speed.Examinees are timed once the first foot passes the acceleration path; the time is stopped once the first foot enters the deceleration path.
Acceleration/deceleration distance for 4mWT at fast speed | 15 minutes
  Distance time that an individual needs to reach their average gait speed. Examinees are timed once the first foot passes the acceleration path; the time is stopped once the first foot enters the deceleration path.

SECONDARY OUTCOMES:
Gait speed for 6mWT | 15 minutes
  Gait speed is the time one takes to walk a specified distance on level surfaces over a short distance.
Gait speed for 4mWT | 15 minutes
  Gait speed is the time one takes to walk a specified distance on level surfaces over a

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Cabanas-Valdés, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richards CL, Malouin F, Dean C. Gait in stroke: assessment and rehabilitation. Clin Geriatr Med. 1999 Nov;15(4):833-55. PMID 10499938
- [Background] Eng JJ, Tang PF. Gait training strategies to optimize walking ability in people with stroke: a synthesis of the evidence. Expert Rev Neurother. 2007 Oct;7(10):1417-36. doi: 10.1586/14737175.7.10.1417. PMID 17939776
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Recovery of walking function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 Jan;76(1):27-32. doi: 10.1016/s0003-9993(95)80038-7. PMID 7811170
- [Background] Geyh S, Cieza A, Schouten J, Dickson H, Frommelt P, Omar Z, Kostanjsek N, Ring H, Stucki G. ICF Core Sets for stroke. J Rehabil Med. 2004 Jul;(44 Suppl):135-41. doi: 10.1080/16501960410016776. PMID 15370761
- [Background] Parker CJ, Gladman JR, Drummond AE. The role of leisure in stroke rehabilitation. Disabil Rehabil. 1997 Jan;19(1):1-5. doi: 10.3109/09638289709166438. PMID 9021278
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Awad L, Reisman D, Binder-Macleod S. Distance-Induced Changes in Walking Speed After Stroke: Relationship to Community Walking Activity. J Neurol Phys Ther. 2019 Oct;43(4):220-223. doi: 10.1097/NPT.0000000000000293. PMID 31449180
- [Background] Montero-Odasso M, Schapira M, Soriano ER, Varela M, Kaplan R, Camera LA, Mayorga LM. Gait velocity as a single predictor of adverse events in healthy seniors aged 75 years and older. J Gerontol A Biol Sci Med Sci. 2005 Oct;60(10):1304-9. doi: 10.1093/gerona/60.10.1304. PMID 16282564
- [Background] Feld JA, Rabadi MH, Blau AD, Jordan BD. Berg balance scale and outcome measures in acquired brain injury. Neurorehabil Neural Repair. 2001;15(3):239-44. doi: 10.1177/154596830101500312. PMID 11944746
- [Background] Taylor-Piliae RE, Latt LD, Hepworth JT, Coull BM. Predictors of gait velocity among community-dwelling stroke survivors. Gait Posture. 2012 Mar;35(3):395-9. doi: 10.1016/j.gaitpost.2011.10.358. Epub 2011 Nov 26. PMID 22119886
- [Background] Cabanas-Valdes R, Garcia-Rueda L, Salgueiro C, Perez-Bellmunt A, Rodriguez-Sanz J, Lopez-de-Celis C. Assessment of the 4-meter walk test test-retest reliability and concurrent validity and its correlation with the five sit-to-stand test in chronic ambulatory stroke survivors. Gait Posture. 2023 Mar;101:8-13. doi: 10.1016/j.gaitpost.2023.01.014. Epub 2023 Jan 20. PMID 36696822
- [Background] Ng SS, Au KK, Chan EL, Chan DO, Keung GM, Lee JK, Kwong PW, Tam EW, Fong SS. Effect of acceleration and deceleration distance on the walking speed of people with chronic stroke. J Rehabil Med. 2016 Oct 5;48(8):666-670. doi: 10.2340/16501977-2124. PMID 27534654
- [Background] Salbach NM, MacKay-Lyons M, Howe JA, McDonald A, Solomon P, Bayley MT, McEwen S, Nelson M, Bulmer B, Lovasi GS. Assessment of Walking Speed and Distance Post-Stroke Increases After Providing a Theory-Based Toolkit. J Neurol Phys Ther. 2022 Oct 1;46(4):251-259. doi: 10.1097/NPT.0000000000000406. Epub 2022 Jun 7. PMID 35671402